CLINICAL TRIAL: NCT01712802
Title: Multicenter Randomized Clinical Study of Denture Adhesive to Establish the Guideline
Brief Title: Multicenter Study of Denture Adhesive
Acronym: DAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nihon University (Other)
Collaborators: Iwate Medical University (Other); Tohoku University (Other); Tsurumi University (Other); Kanagawa Dental University Junior College (Other); Tokyo Medical and Dental University (Other); Osaka Dental University (Unknown); Hiroshima University (Other); University of Tokushima (Other); Nagasaki University (Other); Kagoshima University (Other)
Responsible Party: Principal Investigator, Yasuhiko Kawai, Professor, Nihon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAKEN-24390439
Record Dates: First submitted 2012-10-17; First posted 2012-10-24 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Edentulous
MeSH Terms: conditions — Mouth, Edentulous | interventions — Polident; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Denture Adhesives: Cream (Experimental): Parallel arm that receives application of Cream denture adhesives.
  Interventions: Other: Denture Adhesives: Cream
- Denture Adhesives: Powder (Experimental): Parallel arm that receives application of powder denture adhesive.
  Interventions: Other: Denture Adhesives: Powder
- control (Placebo Comparator): Parallel arm that receive placebo.
  Interventions: Other: Saline

INTERVENTIONS:
Other: Denture Adhesives: Cream — Using Polident as denture adhesive to compare its effect on PRO and subjective outcomes.
  Other Names: Polident
  Arms: Denture Adhesives: Cream
Other: Denture Adhesives: Powder — Using Poligrip powder as denture adhesive to compare its effect on PRO and subjective outcomes.
  Other Names: Poligrip powder
  Arms: Denture Adhesives: Powder
Other: Saline — work as control for Denture Adhesives: Cream and Powder
  Other Names: Otsuka normal saline
  Arms: control

SUMMARY:
To establish evidence based guidelines for denture adhesives (powder and cream), multicenter cross over randomized clinical trial will be carried out.

The null hypotheses are that there are no difference on improvement from baseline to post application of two adhesives powder and cream, in terms of general satisfaction, oral related quality of life, masticatory function and oral conditions.

DETAILED DESCRIPTION:
This is multicenter study of 10 academic affiliated institutions. The clinical trial will be carried out in randomized allocation at each site, and data will be gathered. The intervention will be 3-arms and center institution (Nihon University) will generate each site random numbers for allocation and each site will follow this randomization. Research protocol had been published at Nihon University and distributed to each site.To survey its protocol compliance, the study meeting will be held periodically (twice an year).

ELIGIBILITY:
Inclusion Criteria:

* edentulous

Exclusion Criteria:

* Cannot answer the questionnaire
* Deteriorating general conditions
* Maxillofacial defect
* Metal denture user
* Already denture adhesive users
* Severe xerostomia

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
General satisfaction Patient reported outcomes | day 3 of adhesives application
  General satisfaction (100mm visual analogue scale)

SECONDARY OUTCOMES:
Moisture Objective outcomes | day 3 of each adhesives application
  moisture(%)
masticatory function | day 3 of each adhesives application
  Color change of chewing gum measured by color sensing machine (color scale: categorical)
retentive force | day 3 of each adhesives application
  The maximum occlusal force that can bite before denture moves(N)
Oral related quality of life | day 3 of adhesives application
  Oral health impact profile (OHIP) edentulous Japanese version

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Kawai, DDS MSc PhD, Study Chair — Nihon University
Locations (1):
- Nihon University, Matsudo, Chiba, Japan

REFERENCES:
- [Derived] Ohwada G, Minakuchi S, Sato Y, Kondo H, Nomura T, Tsuboi A, Hong G, Itoh Y, Kawai Y, Kimoto S, Gunji A, Suzuki A, Suzuki T, Kimoto K, Hoshi N, Saita M, Yoneyama Y, Sato Y, Morokuma M, Okazaki J, Maeda T, Nakai K, Ichikawa T, Nagao K, Fujimoto K, Murata H, Kurogi T, Yoshida K, Nishimura M, Nishi Y, Murakami M, Hosoi T, Hamada T. Subjective Evaluation of Denture Adhesives: A Multicenter Randomized Controlled Trial. JDR Clin Trans Res. 2020 Jan;5(1):50-61. doi: 10.1177/2380084419837607. Epub 2019 Apr 11. PMID 30975019
- [Derived] Kimoto S, Kawai Y, Gunji A, Kondo H, Nomura T, Murakami T, Tsuboi A, Hong G, Minakuchi S, Sato Y, Ohwada G, Suzuki T, Kimoto K, Hoshi N, Saita M, Yoneyama Y, Sato Y, Morokuma M, Okazaki J, Maeda T, Nakai K, Ichikawa T, Nagao K, Fujimoto K, Murata H, Kurogi T, Yoshida K, Nishimura M, Nishi Y, Murakami M, Hosoi T, Hamada T. Study protocol for a multi-center, randomized controlled trial to develop Japanese denture adhesive guidelines for patients with complete dentures: the Denture Adhesive Guideline trial: study protocol for a randomized controlled trial. Trials. 2016 Oct 18;17(1):506. doi: 10.1186/s13063-016-1612-x. PMID 27756441